CLINICAL TRIAL: NCT07077226
Title: Prevalence and Clinical Impact of Sleep-Disordered Breathing in Children With Cerebral Palsy at Increased Risk of Respiratory Disorders
Brief Title: Sleep-Disordered Breathing in Children With Cerebral Palsy at Increased Risk of Respiratory Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: GUIDO CAMANNI (Other)
Responsible Party: Sponsor-Investigator, GUIDO CAMANNI, Medical Doctor, Istituto Serafico per sordomuti e per ciechi
Organization: Istituto Serafico per sordomuti e per ciechi (Other)
Other Study IDs: DRSPCI25
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Sleep-disordered Breathing (SDB)
Keywords: sleep-disordered breathing; cerebral palsy; Polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes; Cerebral Palsy | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children (0-17 years) with cerebral palsy who had a sleep study at an Italian reference Center.: Children (0-17 years) of either sex, diagnosed with cerebral palsy who had a sleep study (polysomnography or polygraphy) at an Italian Center during the period 01/01/2020 - 12/31/2023.
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Sleep studies (polysomnography and polygraphy) will be performed and reported according to current American Academy of Sleep Medicine guidelines

SUMMARY:
Currently, there are few and qualitatively unsatisfactory epidemiological data on the prevalence of sleep-disordered breathing (SDB) in children with cerebral palsy (CP).

The investigators aim to conduct a multicentre retrospective study to assess the presence of SDB in children with CP undergoing sleep studies (polysomnography or polygraphy).

DETAILED DESCRIPTION:
A recent review of the scientific literature shows that in the 61 studies on sleep-disordered breathing (SDB) in children with cerebral palsy (CP), epidemiological data on the diagnosis of SDB are scarce and of unsatisfactory quality, as the data are mainly based on the use of targeted questionnaires such as the Pediatric Sleep Questionnaire (PSQ). A study published by Garcia in Developmental Medicine and Child Neurology in 2016 shows that children with CP, especially if they have epilepsy as a comorbidity, have a higher risk of SDB than healthy children.

In a study published in the Annals of Indian Academy of Neurology in 2013, Elsayed found that children with CP are at higher risk for SDB with increasing age, with a higher incidence in the school-age group than in the preschool age group. In the same study, the investigator observed a direct correlation between the severity of motor impairment (levels IV and V versus levels I - III of the Gross Motor Function Classification System scale, GMFCS) and the risk of SDB.

Dum found in 2023 in the Journal of Child Neurology a 2.91-fold (p < 0.001) increased risk of SDB in obese individuals with CP compared to normal weight individuals with CP.

In a retrospective study published in Sleep and Breathing in 2024, Kalyoncu showed good sensitivity (88.8%) of the PSQ in patients with CP, but unacceptable specificity of this instrument (30.7%) compared to polysomnography.

The primary objective of the proposed multicentre retrospective study is to assess the prevalence of SDB in children with diagnosed CP and suspected SDB who underwent polygraphic or polysomnographic examination in the period from 01/01/2020 to 12/31/2023.

A secondary objective is to assess the correlation between SDB and clinical outcome in cases where a follow-up of at least 12 months is available.

Data collected anonymously include clinical aspects (age, gender, GMFCS score, epilepsy diagnosis, adenotonsillar hypertrophy, previous adenotonsillar hypertrophy surgery, spinal changes, previous spinal surgery, oxygen therapy at home, use of Non-Invasive Ventilation/Continuous Positive Airway Pressure (NIV/CPAP) at home, presence of tracheostomy, reported snoring, reported findings of sleep apnea, Assessment of Complex Clinical-Assistance Needs in Pediatrics (ACCAPED) score, referral to a regional palliative care centre) and instrumental (evidence of obstructive sleep apnea in the final diagnosis, mean and minimum oxygen saturation (SPO2), percentage of time with SPO2 <90%, Apnea-Hypopnea Index (AHI), Mixed and Obstructive Apnea-Hypopnea Index (MOAHI), Central Apnea-Hypopnea Index (CAHI), Oxygen Desaturation Index (ODI), heart rate changes).

The following data is collected for the 12-month follow-up after the sleep study: deaths, number of emergency room visits or hospitalisations due to breathing problems, initiation of NIV/CPAP, surgery for adenotonsillar hypertrophy, tracheostomy packing.

ELIGIBILITY:
Inclusion Criteria:

* Aged less than 18 at the time of the sleep study
* A diagnosis of Cerebral palsy
* Written informed consent
* Underwent a sleep study at one of the centers participating in the study during the reporting period (January 2020-December 2023)

Exclusion Criteria:

* None

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children (0-17 years) with cerebral palsy who underwent a sleep study (polysomnography or polygraphy) at one of the Italian centers participating in the study during the period from January 2020 to December 2023
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with obstructive sleep apnea in the study group | The primary outcome measure refers to the first or only sleep study performed by participants in the time interval between January 2020 and December 2023.
  According to the American Academy of Sleep Medicine (AASM), pediatric obstructive sleep apnea (OSA) is diagnosed and classified based on the Apnea-Hypopnea Index (AHI) in the sleep study (polysomnography or polygraphy), which quantifies the number of apnea and hypopnea events per hour of sleep. The sleep study is diagnosed:
  Normal if AHI < 1 event per hour; Mild OSA if AHI is between 1 and 5 events per hour; Moderate OSA if AHI is between 5 and 10 events per hour and Severe OSA if AHI is greater than 10 events per hour.

CONTACTS AND LOCATIONS:
Overall Officials: LUIGI MASINI, MD, Study Chair — OSPEDALE UMBERTO I, SALERNO
Locations (9):
- Italy (9):
  - Uoc Hospice Pediatrico - Azienda Ospedale-Universita' Padova, Padua, PD
  - Uoc Pronto Soccorso Pediatrico Azienda Ospedale-Universita' Padova, Padua, PD
  - Istituto Serafico Di Assisi, Assisi, PG
  - Ospedale Pediatrico Bambino Gesu', Roma, RM
  - Azienda Sanitario-Universitaria Sant'Andrea, Roma, RM
  - Ospedale Umberto I, Salerno, SA
  - Irccs Materno Infantile Burlo Garofolo, Trieste, TS
  - Universita' Degli Studi Dell'Insubria, Varese, VR
  - Azienda Sanitario-Universitaria Federico Ii, Napoli

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol
Time Frame: IPD will be made available for a period of 5 years after completion of the study.
Access Criteria: Substantiated applications for IPD from interested researchers should be sent by e-mail to the sponsor-investigator.

REFERENCES:
- [Background] Kalyoncu M, Namli N, Yegit CY, Yanaz M, Gulieva A, Ergenekon AP, Selcuk M, Atag E, Ikizoglu NB, Sabanci M, Lale K, Gokdemir Y, Ersu R, Karakoc F, Karadag B, Eralp EE. Is the Pediatric Sleep Questionnaire sensitive for sleep-disordered breathing in children with complex chronic disease? Sleep Breath. 2024 Mar;28(1):331-337. doi: 10.1007/s11325-023-02915-z. Epub 2023 Sep 21. PMID 37733254
- [Background] Garcia J, Wical B, Wical W, Schaffer L, Wical T, Wendorf H, Roiko S. Obstructive sleep apnea in children with cerebral palsy and epilepsy. Dev Med Child Neurol. 2016 Oct;58(10):1057-62. doi: 10.1111/dmcn.13091. Epub 2016 Mar 16. PMID 26991829
- [Background] Dum R, Walter V, Thomas NJ, Krawiec C. Odds of Cardiometabolic Diseases and Medications in Children With Cerebral Palsy. J Child Neurol. 2023 Mar;38(3-4):239-246. doi: 10.1177/08830738231167534. Epub 2023 Apr 5. PMID 37016991
- [Background] Elsayed RM, Hasanein BM, Sayyah HE, El-Auoty MM, Tharwat N, Belal TM. Sleep assessment of children with cerebral palsy: Using validated sleep questionnaire. Ann Indian Acad Neurol. 2013 Jan;16(1):62-5. doi: 10.4103/0972-2327.107708. PMID 23661965